CLINICAL TRIAL: NCT06399471
Title: Personalizing MPK Prescription for Individuals With Transfemoral Amputation
Brief Title: Personalizing MPK Prescription
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Kinsey Herrin, Senior Research Scientist, Georgia Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H21008; W81XWH-21-1-0686 (Other Grant/Funding Number: Department of Defense Congressionally Directed Medical Research Program)
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Transfemoral Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Microprocessor Prosthetic Knee (Experimental): Randomization to C-Leg 4.0, Rheo Knee and Power Knee
  Interventions: Device: Microprocessor prosthetic knee

INTERVENTIONS:
Device: Microprocessor prosthetic knee — Microprocessor prosthetic knees for use in a transfemoral prosthesis
  Other Names: C-Leg; Power Knee; Rheo

SUMMARY:
In current clinical prosthetic practice, there is no evidence based method for selecting a microprocessor knee (MPK) joint for a patient with an above the knee amputation. Of individuals with amputation in veteran and service member populations, approximately 35% present with an above the knee amputation. It is well understood in clinical practice that MPKs provide numerous benefits to patients with amputations above the knee including improved gait, safety, comfort, confidence, reduced falls, balance, patient satisfaction and reduced energy expenditure, greater ease in negotiating varying terrains, improvements in multi-tasking and cost effectiveness. Studies that have investigated commercially available MPKs tend to lump all of them together within a single group rather than teasing out individual differences between each knee. Therefore, clinicians are left to rely on their own intuition and past experiences with an MPK when selecting for a patient with an above the knee amputation rather than making their decision based on evidence collected from the specific patient. This may mean that some individuals with an above the knee amputation may not be receiving the best component for them which may delay or inhibit their rehabilitation potential following their amputation.

ELIGIBILITY:
Inclusion Criteria:

* A unilateral transfemoral amputation of the lower limb at least six months post fitting of definitive lower extremity prosthesis
* Habitual use of a lower extremity prosthesis in daily living activities (based on assessment of a physiatrist and/or prosthetist and patient self-report)
* Aged between 18 to 75 years
* K3 or K4 level ambulators who can perform all locomotor tasks of interest (based on assessment of a physiatrist and/or prosthetist)

Exclusion Criteria:

* Individuals with any significant neuromuscular or musculoskeletal disorder or other comorbidity that would interfere with participation (based on assessment of the physiatrist and/or prosthetist and patient self-report)
* Individuals who have open wounds on their residual limb
* Individuals with known visual impairments that would prevent them from safely operating a prosthesis during over ground walking or ascending stairs (based on assessment of the physiatrist and/or prosthetist and patient self-report)
* Individuals with known hearing impairments or who use hearing aids that would prevent them from responding to an auditory instruction (based on assessment of the physiatrist and/or prosthetist and patient self-report)
* Individuals who are currently pregnant (based on patient self-report) due to slight risk of falling during experiments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia Institute of Technology, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herrin K, Kestur S, Zhou S, O'Sullivan G, Snow T, Childers WL, Young A. Toward personalizing prosthesis prescription: A take-home study of three microprocessor-controlled prosthetic knees: A randomized crossover study. PM R. 2025 Oct 24. doi: 10.1002/pmrj.70028. Online ahead of print. PMID 41133928

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Knee condition order was randomized prior to enrollment.
Units Other Than Participants: Prosthetic Knee
Groups:
- Prosthetic Knee Randomized: Each participant performed study activities while wearing a prosthetic knee for one week, followed by a different knee for the second week, and finally a third knee for the third week. The participants in this study have a unilateral transfemoral amputation (i.e. one of their legs is amputated above the knee) and each participant uses a prosthesis to walk. Each participant wore all three knees and were randomized as to which knee they wore on which week. The three knees worn were the Ottobock C-Leg 4.0, Ossur Rheo, and Ossur Power Knee.
Period: Overall Study
Arm/Group | Prosthetic Knee Randomized
Started | 11; 31 Prosthetic Knee
Ottobock C-Leg 4.0 | 10; 10 Prosthetic Knee
Ossur Power Knee | 11; 11 Prosthetic Knee
Ossur Rheo | 10; 10 Prosthetic Knee
Completed | 10; 30 Prosthetic Knee
Not Completed | 1; 1 Prosthetic Knee
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Microprocessor Prosthetic Knee
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: Meters] | 1.75 (0.11)
Weight [Mean (Standard Deviation); unit: Kilograms] | 82.5 (16.3)
AMPnoPro [Mean (Standard Deviation); unit: units on a scale] — The Amputee Mobility Assessment Tool with no Prothesis tool (AMPnoPro) is a 20 item objective measure to characterize mobility. Range is 0 to 43, whereas the higher the score, the more mobility observed. Population: Data was not collected from the one participant who did not complete the study.
  units on a scale
    number analyzed (Participants) | 10
    (all) | 38.1 (3.9)
Clinically Prescribed Prosthetic Knee [Count of Participants; unit: Participants] — Current clinically prescribed knee used in everyday prosthesis.
  Participants
    Otto Bock C-Leg | 7
    Otto Bock X3 | 1
    Plie | 2
    Proteor Quattro | 1

OUTCOME MEASURES:

1. Primary Outcome: Ten Meter Walking Test
Description: Self selected walking speed over ten meters of walking over ground.
Time Frame: 1 month
Population: 1 participant did not complete any of the conditions due to self withdrawal after consenting.
  Each participant wore all three knees during this trial.
Measure: Mean (Standard Deviation); unit: Meters per second
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Meters per second
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 0.9963 (0.2061)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 1.1051 (0.2081)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 1.1111 (0.201)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Power Knee and the C-Leg 4.0 when used during Ten Meter Walking Test; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.126, ANOVA — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary
Statistical Analysis 2: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Power Knee and the Rheo when used during Ten Meter Walking Test; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.015, ANOVA
Statistical Analysis 3: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Rheo and the C-Leg 4.0 when used during Ten Meter Walking Test; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.852, ANOVA

2. Primary Outcome: Two Minute Walking Test
Description: Self selected walking speed over two minutes of walking over ground.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters per second
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Meters per second
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 1.073 (0.2415)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 1.2106 (0.2025)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 1.1698 (0.2458)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Power Knee and the C-Leg 4.0 when used during Two Meter Walking Test; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.003, ANOVA
Statistical Analysis 2: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Power Knee and the Rheo when used during Two Meter Walking Test; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.027, ANOVA
Statistical Analysis 3: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Rheo and the C-Leg 4.0 when used during Two Meter Walking Test; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.425, ANOVA

3. Primary Outcome: Prosthetic Evaluation Questionnaire (PEQ)
Description: A patient reported survey on perceptions of a prosthesis. Scores range zero to one hundred with zero being representing a negative patient reported outcome and one hundred representing a positive patient reported outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
units on a scale
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 69.4 (8.99)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 83.2 (10.15)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 78.4 (11.75)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; The Non-parametric Friedman's test was used to compare the survey results between the participants using the Power Knee and the C-Leg 4.0; Test type: Other — Non-parametric Friedman's test with multiple comparison correction; p = 0.006, Non-parametric Friedman's test with mult
Statistical Analysis 2: Comparison: Prosthetic Knee Randomized; The Non-parametric Friedman's test was used to compare the survey results between the participants using the Power Knee and the Rheo; Test type: Other — Non-parametric Friedman's test with multiple comparison correction; p = 0.236, Non-parametric Friedman's test with mult
Statistical Analysis 3: Comparison: Prosthetic Knee Randomized; The Non-parametric Friedman's test was used to compare the survey results between the participants using the Rheo and the C-Leg 4.0; Test type: Other — Non-parametric Friedman's test with multiple comparison correction; p = 0.118, Non-parametric Friedman's test with mult

4. Secondary Outcome: Stance Time Asymmetry Index
Description: Stance time asymmetry index measures the percent difference in stance time between the prosthetic and sound side limbs. A value equal to zero is indicative of perfect symmetry. Negative values of ST asymmetry index are indicative of increased time spent on the sound side and positive values are indicative of increased time on the prosthetic side.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of stance time
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
percentage of stance time
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | -10.15 (3.68)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | -10.95 (9.98)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | -7.03 (8.13)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Power Knee, the C-Leg 4.0, and the Rheo when used during Stance Time Asymmetry Index test; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.687, ANOVA

5. Secondary Outcome: Narrowing Beam Walking Test
Description: A measure of balance via walking down a narrowing beam.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Feet
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Feet
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 11.3 (3.14)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 12.6 (2.80)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 13.5 (2.64)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Power Knee, the C-Leg 4.0, and Rheo when used during the Narrowing beam walking test; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.082, ANOVA

6. Secondary Outcome: Reported Falls
Description: Average reported falls per day.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Falls per day
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Falls per day
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 0.06429 (0.10326)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 0.04286 (0.06547)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 0.01429 (0.04286)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the reported falls when for when the Power Knee, C-Leg 4.0, and the Rheo were used; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.943, ANOVA

7. Secondary Outcome: Physiological Cost Index
Description: A clinical measure of energy expenditure. This formula consists of working heart minus resting heart rate divided by speed.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Heart beats per meter
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Heart beats per meter
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 0.29 (0.1034)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 0.25 (0.0593)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 0.27 (0.0984)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Physiological cost index for when the Power Knee, the C-Leg 4.0, and the Rheo were used; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.535, ANOVA

8. Secondary Outcome: Stair Ascent Speed
Description: Self selected walking speed during stair ascent.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Steps per minute
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Steps per minute
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 50.463 (7.9767)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 56.336 (17.494)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 48.336 (7.1067)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Stair Ascent Speed for the Power Knee, C-Leg 4.0, and the Rheo when used; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.229, ANOVA

9. Secondary Outcome: Stair Descent Speed
Description: Self selected walking speed while descending stairs.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Steps per minute
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Steps per minute
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 92.65 (25.67)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 93.997 (27.183)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 88.3 (21.261)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Stair Descent Speed for the Power Knee, C-Leg 4.0, and the Rheo when used; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.528, ANOVA

10. Secondary Outcome: Ramp Ascent Speed
Description: Self selected walking speed while ascending a 5 degree incline.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters per second
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Meters per second
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 0.8929 (0.1533)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 0.969 (0.2086)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 0.971 (0.1754)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Ramp Ascent Speed between the Power Knee and the C-Leg 4.0; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.144, ANOVA
Statistical Analysis 2: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Ramp Ascent Speed between the Power Knee and the Rheo; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.024, ANOVA
Statistical Analysis 3: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Ramp Ascent Speed between the Rheo and the C-Leg 4.0; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.949, ANOVA

11. Secondary Outcome: Ramp Descent Speed
Description: Self selected walking speed while descending a 5 degree incline.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters per second
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 10
Number analyzed (Prosthetic Knees) | 30
Meters per second
  Power Knee: number analyzed (Prosthetic Knees) | 10
  Power Knee | 0.7643 (0.1675)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 10
  C-Leg 4.0 | 0.869 (0.2282)
  Rheo: number analyzed (Prosthetic Knees) | 10
  Rheo | 0.8584 (0.2436)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Ramp Descent Speed for the Power Knee, C-Leg 4.0, and the Rheo when used; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.051, ANOVA

12. Secondary Outcome: Steps Per Day
Description: Steps per day as measured by StepWatch.
Time Frame: 1 month
Population: 1 participant did not complete any of the conditions due to self withdrawal after consenting.
  No data obtained from two participants due to experimental error.
  Each participant wore all three knees during this trial.
Measure: Mean (Standard Deviation); unit: Steps per day
Units Other Than Participants: Prosthetic Knees
Arm/Group | Prosthetic Knee Randomized
Number analyzed (Participants) | 8
Number analyzed (Prosthetic Knees) | 24
Steps per day
  Power Knee: number analyzed (Prosthetic Knees) | 8
  Power Knee | 2620.1 (705.5)
  C-Leg 4.0: number analyzed (Prosthetic Knees) | 8
  C-Leg 4.0 | 2762.6 (969.2)
  Rheo: number analyzed (Prosthetic Knees) | 8
  Rheo | 2462.6 (1030.2)
Statistical Analysis 1: Comparison: Prosthetic Knee Randomized; An ANOVA was used to compare the Steps per Day for the Power Knee, C-Leg 4.0, and the Rheo when used; Test type: Other — One-way Repeated Measures ANOVA with sphericity correction (Huynh-Feldt) applied if necessary; p = 0.367, ANOVA

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Ottobock C-Leg 4.0: Each participant performed study activities while wearing the Ottobock C-Leg 4.0 prosthetic knee for one week. The participants in this study have a unilateral transfemoral amputation (i.e. one of their legs is amputated above the knee) and each participant uses a prosthesis to walk.
- Ossur Rheo: Each participant performed study activities while wearing the Ossur Rheo prosthetic knee for one week. The participants in this study have a unilateral transfemoral amputation (i.e. one of their legs is amputated above the knee) and each participant uses a prosthesis to walk.
- Ossur Power Knee: Each participant performed study activities while wearing the Ossur Power Knee prosthetic knee for one week. The participants in this study have a unilateral transfemoral amputation (i.e. one of their legs is amputated above the knee) and each participant uses a prosthesis to walk.
Arm/Group | Ottobock C-Leg 4.0 | Ossur Rheo | Ossur Power Knee
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT06399471/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT06399471/ICF_001.pdf